CLINICAL TRIAL: NCT01578278
Title: Bepotastine Besilate-corticosteroid Nasal Spray Combination Compared to Placebo, Bepotastine Besilate Nasal Spray, and Corticosteroid Nasal Spray in the Treatment of Patients With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S00186
Record Dates: First submitted 2012-01-18; First posted 2012-04-16 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Bepotastine besilate formulation (Experimental): Nasal Spray
  Interventions: Drug: Bepotastine besilate formulation
- Fluticasone propionate (Experimental): Nasal Spray
  Interventions: Drug: Fluticasone propionate
- Bepotastine besilate-fluticasone propionate (Experimental): Nasal Spray
  Interventions: Drug: Bepotastine besilate-fluticasone propionate
- Placebo Comparator (Placebo Comparator): Nasal Spray
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Bepotastine besilate formulation — Nasal Spray
  Arms: Bepotastine besilate formulation
Drug: Fluticasone propionate — Nasal Spray
  Arms: Fluticasone propionate
Drug: Bepotastine besilate-fluticasone propionate — Nasal Spray
  Arms: Bepotastine besilate-fluticasone propionate
Drug: Placebo Comparator — Nasal Spray
  Arms: Placebo Comparator

SUMMARY:
This is a clinical study to evaluate the safety and efficacy of a bepotastine besilate-corticosteroid combination nasal spray for the treatment of seasonal allergic rhinitis (SAR) in an open exposure study with subjects who have a demonstrated history of Mountain Cedar pollen allergy. The primary study objective is to assess the reduction from baseline in averaged morning (AM) and evening (PM) values of reflective total nasal symptom scores for each of 3 nasal sprays (bepotastine besilate-fluticasone propionate combination nasal spray, bepotastine besilate nasal spray, fluticasone propionate nasal spray) compared to placebo nasal spray. For enrolled subjects, the study will involve a 7-10 day run-in screening period dosing with placebo nasal spray and then a 14-day treatment period where subjects will dose twice a day with 1 of the 4 test agent nasal sprays and record reflective and instantaneous scores for both nasal and ocular symptoms prior to each dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 12 years of age with a demonstrated history of Mountain Cedar pollen allergy

Exclusion Criteria:

* No active nasal infection or nasal abnormality that would affect subject safety or symptom assessments

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bepotastine Besilate-fluticasone Propionate: Nasal Spray
  Bepotastine besilate 4%-fluticasone propionate 0.05%: Nasal Spray
- Bepotastine Besilate Formulation: Nasal Spray
  Bepotastine besilate formulation 4%: Nasal Spray
- Fluticasone Propionate: Nasal Spray
  Fluticasone propionate 0.05%: Nasal Spray
Period: Overall Study
Arm/Group | Bepotastine Besilate-fluticasone Propionate | Bepotastine Besilate Formulation | Fluticasone Propionate | Placebo Comparator
Started | 152 | 152 | 154 | 148
Completed | 148 | 150 | 150 | 139
Not Completed | 4 | 2 | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bepotastine Besilate-fluticasone Propionate | Bepotastine Besilate Formulation | Fluticasone Propionate | Placebo Comparator | Total
Number analyzed (Participants) | 152 | 152 | 154 | 148 | 606
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (14.8) | 43.4 (14.4) | 40.6 (14.8) | 43.6 (13.9) | 41.4 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 95 | 89 | 89 | 383
  Male | 42 | 57 | 65 | 59 | 223

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (Pre-Dose) in Morning and Evening Averaged Subject-rated Reflective TNSS
Description: Total nasal symptom scores (TNSS) was the summed scores for nasal pruritus [itching], rhinorrhea [runny nose], nasal congestion, and sneezing. Individual nasal symptoms were rated on a 4-point scale from 0-3 (0=Absent, 1=Mild, 2=Moderate, 3=Severe), with no half-unit assessments. TNSS was the sum score of 4 nasal symptoms with a minimum score of 0 and a maximum score of 12 units, with higher score corresponding to increased severity of nasal allergy symptoms. The morning and evening scores were averaged.
Time Frame: Baseline, 14 days
Population: All randomized participants were included in the analysis population, with last observation carried forward used for missing data at 14 days.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bepotastine Besilate-fluticasone Propionate | Bepotastine Besilate Formulation | Fluticasone Propionate | Placebo Comparator
Number analyzed (Participants) | 152 | 152 | 154 | 148
score on a scale | -3.57 (2.82) | -2.31 (2.43) | -2.96 (2.73) | -1.48 (1.99)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Bepotastine Besilate-fluticasone Propionate | Bepotastine Besilate Formulation | Fluticasone Propionate | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/152 | 0/154 | 0/148
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/152 | 0/154 | 0/148
Other Adverse Events (participants affected / at risk) | 9/152 | 8/152 | 0/154 | 0/148
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bepotastine Besilate-fluticasone Propionate (N=152) | Bepotastine Besilate Formulation (N=152) | Fluticasone Propionate (N=154) | Placebo Comparator (N=148)
Mild taste following instillation (General disorders) | 9 | 8 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.